CLINICAL TRIAL: NCT06996236
Title: Brimonidine Eye Drops in the Prevention of Myopia Progression
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fundacion para la Investigacion Biomedica del Hospital Universitario Ramon y Cajal (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: BPM2024
Record Dates: First submitted 2025-04-22; First posted 2025-05-30 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lumobry 0.25 mg/ml eye drops solution (Active Comparator): Lumobry 0.25 mg/ml eye drops solution
  Interventions: Drug: Treatment with brimonidine eye drops 0.025%

INTERVENTIONS:
Drug: Treatment with brimonidine eye drops 0.025% — Treatment with brimonidine eye drops 0.025%, instilled once a day at night, with simultaneous occlusion of the lower lacrimal punctum to avoid its systemic absorption, for 2 years.

SUMMARY:
Study to determine the efficacy of alpha-2 adrenergic drugs (brimonidine) in the prevention of myopia progression. Given that the drugs used so far have limited efficacy and side effects (loss of near vision, photophobia), it may be an interesting contribution to such treatment at low cost, and to avoid the expense of managing the complications of myopia that develop throughout life.

DETAILED DESCRIPTION:
For the prevention of myopia progression it is reasonable to use a local topical route in eye drops, since it avoids the occurrence of systemic side effects and the drug reaches the corresponding receptors at a higher concentration via the topical route. This route of administration has been previously used in animal models and in humans, with atropine, pirenzepine and brimonidine.

The concentration proposed (0.025%) in this study is the one used with relative success without side effects for atropine in humans, and has also been used in animal models for brimonidine itself. As this is a first study, the investigators do not propose the use of higher concentrations at this time. The proposed regimen (once a day) is the one commonly used in the treatment of myopia. Although at the concentration used it is used 3-4 times a day in other indications of brimonidine eye drops, given the longer duration of this treatment and the fact that it is a first study, the investigators opted for the once-daily regimen.

Since eye growth is relatively slow, a treatment duration of 1 to 2 years is necessary to assess the effect of the drug on myopia progression and eye axial length variation. In addition, in case of therapeutic use of brimonidine eye drops, it would be necessary to use it for long periods of time, not less than 2 years, so it is convenient to evaluate its behavior when used in long term regimens.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 6 to ≤ 14 years
* Patients who, after having received information about the design, the purposes of the study, the possible risks that may arise from it and that at any time they may refuse to cooperate, give written consent to participate in the study (the patient older than 12 years and the legal representative)
* Myopia ≥ -1. 50 Diopters of spherical equivalent, ranging from -1.50 to -5.50 D
* Astigmatism with a cylinder power ≤ -1.50 Diopters
* Anisometropia (refractive difference between both eyes) in spherical equivalent ≤ 1.25 Diopters
* Visual acuity (CVA) > 0.3 logMAR (0.5 on Snellen scale).
* Intraocular pressure < 20 mm Hg
* In women of childbearing age negative urine pregnancy test performed within 7 days prior to the start of treatment
* Women and men with partners of childbearing age must agree to use a highly effective method of contraception (such as surgical sterilization, double barrier method, oral contraceptives or hormonal contraceptive implants) and to continue using them until 6 months after the last dose of treatment.

Exclusion Criteria:

* Presence of any other ocular pathology (other than myopia)
* History of allergy to the medications and excipients used in the study
* History of previous therapy for myopia using eye drops, contact lenses or multifocal or bifocal glasses
* Amblyopia (2 or more lines of difference in visual acuity between both eyes, on logMAR scale, with optical correction)
* Any of the following situations present at the time: prolonged ocular hyperemia, prolonged ocular irritation, ocular infections - mucopurulent discharge in ocular tissues, ocular pain, vision changes/alterations other than myopia
* Any clinical situation that at the investigator's discretion advises against participation.

Ages: 6 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Effect of brimonidine eye drops 0.025% on myopia progression in children aged 6 to 14 years | 24 months
  Progression of myopia (change in spherical equivalent of refractive error) measured every 6 months (Auto-refractometry and Subjective refraction)

SECONDARY OUTCOMES:
Progression of various ocular biometric variables in the children of the treated and control groups, | 24 months
  Myopia progression by measuring every 6 months: change in axial eye length
Progression of various ocular biometric variables in the children of the treated and control groups | 24 months
  Description: Myopia progression by measuring every 6 months: visual acuity
Progression of various ocular biometric variables in the children of the treated and control groups | 24 Months
  Description: Myopia progression by measuring every 6 months: pupillometry/accommodation
Progression of various ocular biometric variables in the children of the treated and control groups | 24 Months
  Description: Myopia progression by measuring every 6 months: corneal topography
Progression of various ocular biometric variables in the children of the treated and control groups | 24 Months
  Description: Myopia progression by measuring every 6 months: intraocular pressure
Progression of various ocular biometric variables in the children of the treated and control groups | 24 Months
  Collecting adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario Ramón y Cajal, Madrid, Madrid, Spain